CLINICAL TRIAL: NCT04596592
Title: Pubertal Blockade and Estradiol Effects on Cardiometabolic Health for Transitioning Youth
Acronym: PUBERTY
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-1226; 1K23HL151868-01 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2020-10-22 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Transgenderism; Gender Dysphoria; Insulin Sensitivity
MeSH Terms: conditions — Transsexualism; Gender Dysphoria; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional consent for DNA collection and storage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender
- Cisgender

SUMMARY:
To evaluate the effect of estradiol with or without a prior gonadotropin releasing hormone analogue on insulin sensitivity and vascular function in transgender females compared to cisgender controls.

ELIGIBILITY:
Inclusion Criteria (transgender females):

* Identify as a transgender female
* Age 13-16 years at the time of enrollment
* If on a gonadotropin releasing hormone analogue, > 6 months exposure
* Plan to start estradiol clinically in < 4 months

Inclusion Criteria (cisgender males and females):

* Males and females ages 13-16 years

Exclusion Criteria:

* Cognitive, psychiatric, or physical impairment resulting in inability to tolerate the study procedures
* Antipsychotic medication use
* Type 1 or 2 diabetes (by medical history)
* Polycystic ovarian syndrome (PCOS for cisgender females)
* Hypertension (resting BP ≥ 140/90 mm/Hg)
* Weight> 400 lbs
* On oral progesterone medications (including oral progesterone or progestin, combined oral contraceptives or etonogestrel implant)
* Pregnancy (for cisgender females)

Ages: 13 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Transgender and cisgender adolescents
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline to 12 months
Brachial artery flow mediated dilation | Change from baseline to 12 months

SECONDARY OUTCOMES:
Large artery stiffness | Change from baseline to 12 months
  Carotid artery ultrasound
Cerebrovascular function | Change from baseline to 12 months
  Middle cerebral artery blood flow
VO2 peak | Change from baseline to 12 months
Fat mass | Change from baseline to 12 months
  DXA
Fat-free mass | Change from baseline to 12 months
  DXA

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Nokoff, MD, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No